CLINICAL TRIAL: NCT04577352
Title: A Randomized, Parallel-Arm, Double-Blind, Placebo-Controlled Study With Open-Label Extension to Assess the Efficacy and Safety of Vatiquinone for the Treatment of Friedreich Ataxia (MOVE-FA)
Brief Title: A Study to Assess the Efficacy and Safety of Vatiquinone for the Treatment of Participants With Friedreich Ataxia
Acronym: MOVE-FA
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: PTC Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PTC743-NEU-003-FA
Record Dates: First submitted 2020-09-30; First posted 2020-10-06 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-03

CONDITIONS: Friedreich Ataxia
MeSH Terms: conditions — Friedreich Ataxia | interventions — alpha-tocotrienol quinone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Vatiquinone (Experimental): Participants will receive vatiquinone capsule at a dose of either 200 milligrams (mg) orally 3 times a day (TID) if ˂12 years of age and weighing ˂25 kilograms (kg) or 400 mg orally TID if ≥12 years of age and/or weighing ≥25 kg for 72 weeks during the placebo-controlled phase and for 24 weeks during the open-label extension phase.
  Interventions: Drug: Vatiquinone
- Placebo (Placebo Comparator): Participants will receive placebo matching to vatiquinone (per age and weight) orally TID for 72 weeks during the placebo-controlled phase and vatiquinone at a dose of either 200 mg orally TID if ˂12 years of age and weighing ˂25 kg or 400 mg orally TID if ≥12 years of age and/or weighing ≥25 kg for 24 weeks during the open-label extension phase.
  Interventions: Drug: Vatiquinone; Drug: Placebo

INTERVENTIONS:
Drug: Vatiquinone — Vatiquinone will be administered per dose and schedule specified in the arm.
Drug: Placebo — Placebo will be administered per schedule specified in the arm.
  Arms: Placebo

SUMMARY:
The primary objective of the study is to evaluate the efficacy (using the modified Friedreich Ataxia Rating Scale [mFARS]) and safety of vatiquinone in participants with Friedreich ataxia (FA).

DETAILED DESCRIPTION:
During the double-blind, placebo-controlled phase, participants will be stratified by baseline mFARS score (<40 versus ≥40), age of disease onset (<14 versus ≥14), and age at screening (≤21 years or >21 years) and randomized to receive either vatiquinone or placebo using interactive response technology (IRT). Following completion of the randomized, double-blind, placebo-controlled phase (72 weeks), participants will enter into an open-label extension phase (24 weeks) during which they will receive open-label treatment with vatiquinone at the dose they received in the randomized phase of the study (for participants entering the extension phase who initially received placebo, the dose of vatiquinone will be determined based on age and weight) and then a safety follow-up (approximately 30 days [±5 days] after last dose or termination visit, whichever is later).

The primary efficacy analysis will be based on change from baseline in mFARS score of participants between 7 and 21 years old. In order to explore the treatment efficacy and safety, approximately an additional 20 participants >21 years of age will be randomized for a total of approximately 126 participants.

ELIGIBILITY:
Inclusion Criteria:

* mFARS ≥20 to ≤70 at baseline
* Must be able to ambulate at least 10 feet in 1 minute with or without assistance (non-wheelchair).
* Friedreich ataxia diagnosis (homozygous for guanine-adenine-adenine [GAA] repeat expansion in intron-1 of frataxin [FXN] gene), confirmed by clinical testing (Note: size of GAA repeat is not required for eligibility)
* Consent to comply with study procedures. For participants under the age of 18 (or age of consent), parent(s)/legal guardian(s) of the participant must agree to comply with the requirements of the study, including the need for frequent and prolonged follow up; parent(s)/legal guardian(s) with custody of the participant must give their consent for participant to enroll in the study.
* Difference in the mFARS at screening and baseline of no more than 4 points.
* Must be able to abstain from anticoagulants and any aspirin (including 81 mg) for 30 days prior to the baseline visit and for the duration of the study; any possible discontinuation of anticoagulants should be monitored and indicated by a specialist (for example, cardiologist, neurologist, or hematologist) and discontinuation will be noted by the prescribing physician.
* Must be able to abstain from potent cytochrome P450 (CYP) 3A4 inducers/inhibitors (for example, ketoconazole, rifampin, St. John's wort, grapefruit juice or any grapefruit product) for at least 30 days prior to enrollment
* Must be able to swallow capsules
* Males and females of childbearing potential must be willing to use an effective method of contraception from the time consent is signed until 30 days after the last dose of study drug or early termination visit. Male participants must agree not to donate sperm during the study and for at least 30 days after the last dose of study drug or early termination visit.

Exclusion Criteria:

* Individuals with clinical diagnosis of FA who have point mutations or deletions or other non-GAA expansion mutations
* Previous treatment with vatiquinone
* Allergy to vatiquinone, sesame oil, gelatin (bovine and/or porcine), titanium dioxide, or red iron oxide
* Ejection fraction <50%
* Uncontrolled diabetes (glycated hemoglobin [HbA1c] >7.0%) at the time of screening
* Has current suicidal ideation based on Columbia-Suicide Severity Rating Scale (C-SSRS) within 3 months prior to screening or between screening and baseline at the baseline visit or suicidal behavior within the last year at the screening visit or between screening and baseline at the baseline visit
* Pregnant or lactating participants or those sexually active participants who are unwilling to comply with proper birth control methods; females of childbearing potential must have a negative pregnancy test at screening and during the baseline visit
* Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) ≥2 * upper limit of normal (ULN) at time of screening
* International normalized ratio (INR) ≥1.5 * ULN at time of screening or clinically significant (CS) bleeding, as determined by the investigator
* Serum creatinine ≥1.5 * ULN at time of screening
* Comorbidities that may confound study results (for example, fat malabsorption syndrome, other mitochondrial disorder) in the opinion of the investigator
* Participation in any other interventional clinical trial or received any investigational drug in any other clinical trial within 60 days prior to the baseline visit. Participants may be rescreened after the exclusionary period of 60 days has passed.
* Concomitant use of interventional coenzyme Q10 (CoQ10), vitamin E, or any approved or non-approved medication for FA within 30 days prior to the screening visit. These prohibited medications can be discontinued at the screening visit; if this is the case, the mFARS assessment must be repeated to confirm inclusion eligibility after a minimum of 30 days post-discontinuation and there must be no more than a 4-point difference in mFARS assessed from the post-discontinuation visit to the baseline visit.
* Illicit drug use 30 days prior to screening and during the study is prohibited.

Min Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2020-12-17 (Actual); Primary Completion 2023-04-04 (Actual); Study Completion 2023-10-02 (Actual)

PRIMARY OUTCOMES:
Change From Baseline in the Modified Friedreich Ataxia Rating Scale (mFARS) Score at Week 72 | Baseline, Week 72
  Friedreich Ataxia Rating Scale (FARS) is a disease-specific scale that measures progression of neurological effects of FA. The mFARS is a validated and reliable 93- item scale; comprised of the neurologic component of the FARS and evaluates bulbar, upper limb, lower limb, and upright stability/gait function. For each item, responses categorize the corresponding neurological finding, and the findings are assigned a score ranging from 0 to 3, 4, or 5 with 0 being normal and higher numbers indicative of greater impairment.

SECONDARY OUTCOMES:
Change From Baseline in Friedreich Ataxia Rating Scale Activities of Daily Living (FARS-ADL) Score at Week 72 | Baseline, Week 72
  The FARS-ADL is a subsection of the FARS questionnaire that assesses activities of daily living, including speech, personal hygiene, feeding, and mobility. Participants rank each category using a scale of 0 (normal) to 4 (severe disability/ inability to carry out activity independently), with lower scores indicative of "normal" function/activity.
Change From Baseline in 1-Minute Walk Test (1MWT) at Week 72 | Baseline, Week 72
  The 1MWT is a timed performance test used to measure functional ability, walking endurance, balance, and muscle performance by measuring maximal walking speed in 1 minute. Participants will be instructed to walk as quickly as possible for 1 minute without running. Maximal walking speed will be measured upon completion of the walk and recorded.
Number of Falls Through Week 72 | Baseline through Week 72
  The fall log directly relate to a participant's ability to ambulate during normal daily activities. Thus, each participant will be required to maintain a fall log, which will include the date and time of each fall. Falls as defined by World Health Organization as "inadvertently coming to rest on the ground, floor or other lower level, excluding intentional change in position to rest in furniture, wall or other objects," will be reported.

CONTACTS AND LOCATIONS:
Locations (14):
- United States (5):
  - UCLA, Los Angeles, California
  - University of Florida, Gainesville, Florida
  - University of South Florida, Tampa, Florida
  - University of Iowa, Iowa City, Iowa
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
- Murdoch Children's Research Institute, Parkville, Victoria, Australia
- University of Campinas (UNICAMP) - School of Medical Sciences, Dept of Neurology, São Paulo, Brazil
- Canada (2):
  - Centre de Recherche du Centre Hospitalier de l'Université de Montreal (CRCHUM), Montreal, Quebec
  - CHU Sainte-Justine, Montreal, Quebec
- Hôpital Pitié-Salpêtrière, Institut du Cerveau (Paris Brain Institute), Paris, France
- Department of Neurology and Hertie-Institute for Clinical Brain Research German Center of Neurodegenerative Diseases (DZNE), Tübingen, Germany
- Ospedale Pediatrico Bambino Gesu' IRCCS, Roma, Italy
- CBR Neurogenetic Research Clinic, University of Auckland, Auckland, New Zealand
- Hospital Sant Joan de Déu Barcelona Unidad de Enfermedades Neuromusculares, Barcelona, Spain